CLINICAL TRIAL: NCT05597592
Title: Experimentation of a Personalized Physical Self-education Program at Home: Feasibility Study (PROSOL TELEKINECT)
Acronym: TELEKINECT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no subcontractors for management of connected watches
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-PP-13
Record Dates: First submitted 2022-10-17; First posted 2022-10-28 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-01

CONDITIONS: Neuromuscular Diseases; Neurodegenerative Diseases
MeSH Terms: conditions — Neuromuscular Diseases; Neurodegenerative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with neuromuscular or neurogenerative disease (Experimental)
  Interventions: Procedure: Feasability of a personalised physical rehabilitation program at home

INTERVENTIONS:
Procedure: Feasability of a personalised physical rehabilitation program at home — Monitoring of the realization of a personalised physical rehabilitation program at home by patients with neuromuscular and neurodegenrative disease

SUMMARY:
ALCOTRA (Alpes Latines COoperation TRAnsfrontalière) is one of the European cross-border cooperation programmes covering France and Italy and financed by the ERDF (European Regional Development Fund). It includes the thematic plan (PITEM), called "PROSOL" (PROximity and SOLidarity), set up in the PIEDMONT region (Italy). The PITEM PROSOL strategy aims to develop new social and health services for vulnerable populations in the rural areas and cross-border Franco-Italian mountains of the South regions (Provence Alpes Cote d'Azur, Liguria, Piedmont and Aosta valley).

As part of the PITEM PROSOL project, a PROSOL telemedicine platform has been developped for the management of isolated patients from the territory of the Latin Alpes and suffering from neurological diseases (neurodevelopmental disorders, neuromuscular diseases and neurodegenerative diseases). These patients are divided into 3 experimental groups: WOMEN (project 5106), SENIORS (project 4128) and YOUTH (project 5162). A PROSOL e-learning platform (https://www.prosol-elearning.com/) has also been developped for these patients, their caregivers and community physicians to improve knowledge and management of these diseases.

Experimentation of these platforms by several participants (and their caregivers) has highlighted the need, often discontent, of a personalized management of physiotherapy for patients with neuromuscular diseases (MNM) and neurodegenerative diseases (Alzheimer's disease). As physical activity has a beneficial and protective effect of these diseases, and inactivity is one of the important risk factors in worsening symptoms contributing to the loss of patients' motor and cognitive functional abilities, a program of self-physical rehabilitation has been designed by neurologists and physiotherapists of expert centers for a personalized and adapted treatment for each patient.

The PROSOL TELEKINECT project offers a physical rehabilitation program to be carried out autonomously at home, with coaching by physiotherapists via the telemedicine platform, as well as close monitoring of exercise response regarding the level of pain and fatigue of patients, thus ensuring their maximum safety.

The objective of the PROSOL TELEKINECT project is to evaluate the value of an appropriate physical rehabilitation programme for each type of patient. The feasibility and beneficial effects of this program will be assessed using conventional assessments of motor function and patient quality of life, but also using a connected watch coupled with artificial intelligence algorithms to collect and analyze physiological data remotely in real time in the patients' natural environment.

The results of this pilot study will be used to lay the foundation for a larger clinical study to test a new digital strategy for self-treatment rehabilitation, aimed at reducing unequal access to care for patients with neuromuscular and neurodegenerative diseases, and residents of transboundary territories, thus offering the establishment of a preventive and supportive approach to these diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age higher than 18 years old
* Patient living in the cross-border region concerned by the PROSOL project (Provence Alpes Cote d'Azur, Liguria, Piedmont and Aosta valley)
* Patient with neuropathy with genetic confirmation or myopathy with genetic confirmation or a minor neurocognitive disorder (DSM V criteria) with a Mini Mental State Examination (MMSE) score greater tha or equal to 15 and less than 26
* Patient able to perform the self-rehabilitation program alone or with the help of a caregiver (at the investigator's discretion): ambulant patients alone or with assistance (group 1) or non-ambulant patients able to transfer independently (group 2)
* Likely to be followed by telemedicine (equipped with a smartphone (Apple or Android) and/or a computer, a camera, an internet connection, the smartphone should be compatible with the use of the connected watch (possibility to download mobile applications: Healthmate, Link4life and Telegram
* Patient not planning any change in his lifestyle in the month following the inclusion (hiking, joining a gym, total immobility...)
* Patient able to comply with the instructions and procedures specified in the clinical protocol
* Patient has given free and informed consent
* Patient affiliated to a social security system.

Exclusion Criteria:

* Patient with balance disorders that are incompatible with the proper conduct of the study based on the investigator's judgment at the inclusion visit
* Patient with any pathologies or comorbidities incompatible with the proper conduct of the study according to the investigator's judgement during the inclusion visit (heart problems, respiratory problems, etc…)
* Patient with pacemaker (this could interfere with data collected by the smartwatch)
* Patient with respiratory problems requiring non-invasive ventilation (NIV) or oxygen therapy
* Patient presenting or having presented in the previous month the inclusion of average physical tiredness (EVA tiredness > 6)
* Patient presenting or having presented in the month before the inclusion of myalgia (EVA pain > 6)
* Pregnant or lactating woman or woman of childbearing age without contraception
* Patient protected by law under guardianship or curatorship, or not able to participate in a clinical study under article L. 1121-16 of the French Public Health Code
* Patient refusing to participate in the study or expressing opposition to participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate feasability of a personalized physical rehabilitation program at home | 4 weeks
  Feasability will be assessed by the number of complete training session performed by each patient. A complete program is composed of 3 sessions per week, during 2 weeks. The program will be considered feasible if at least 80% of patients have completed correctly all the training program.

SECONDARY OUTCOMES:
Evaluate the feasability of measuring the impact of a personalized physical rehabilitation program at home on the daily physical activity at S1, S2, S3 and S4 | one week before the program (S1), 2 weeks of the program (S2 and S3) and one week after the end of the program (S4)
  The daily physical activity will be assessed by the daily distance travelled by ambulant patients. This daily distance will be compared, for each patient, between the week before the program (S1), during the 2 weeks of program (weeks S2 and S3) and the week after the end of the program (S4).
Evaluate the feasability of measuring the impact of a personalized physical rehabilitation program at home on the heart rate, one week before the program (S1) and one week after the end of the program (S4) | one week before the program (S1) and one week after the end of the program (S4)
  Heart rate will be collected every day using a connected watch
Evaluate the feasability of measuring the impact of a personalized physical rehabilitation program at home on electrocardiogram (heart cycle), one week before the program (S1) and one week after the end of the program (S4) | one week before the program (S1) and one week after the end of the program (S4)
  Electrocardiogram will be collected every day using a connected watch. Regularity of heart cycle will be analysed.
Evaluate the feasability of measuring the impact of a personalized physical rehabilitation program at home on electrocardiogram (atrial fibrillation), one week before the program (S1) and one week after the end of the program (S4) | one week before the program (S1) and one week after the end of the program (S4)
  Electrocardiogram will be collected every day using a connected watch. Evidence of atrial fibrillation will be analysed
Evaluate the feasability of measuring the impact of a personalized physical rehabilitation program at home on respiratory function, one week before the program (S1) and one week after the end of the program (S4) | one week before the program (S1) and one week after the end of the program (S4)
  Respiratory function will be assessed by the pulse oxugen saturation (SpO2) collected by the connected watch. Value of SpO2 will be compared between one week before the program (S1) and one week after the end of the program (S4)
Evaluate the feasability of measuring the impact of a personalized physical rehabilitation program at home on quality of life for patients with neuromuscular diseases, at V1 and V3 | At inclusion visit (V1) and at 4 weeks (V3)
  Quality of life of patients with neuromuscular disease will be assessed using the "Individualised Neuromuscular Quality of Life Questionnaire" (INQol, version 2).
Evaluate the feasability of measuring the impact of a personalized physical rehabilitation program at home on quality of life for patients with neurodegenerative diseases, at V1 and V3 | At inclusion visit (V1) and at 4 weeks (V3)
  Quality of life of patients with neuromuscular disease will be assessed using the "The Alzheimer's Disease-Related Quality of Life" (ADRQL).
Evaluate the feasability of measuring the impact of a personalized physical rehabilitation program at home on global felt tiredness, before the program at V1, between S2 and S3 and at V3 | At inclusion visit (V1), between week 2 and 3 (S2 or S3) and at 4 weeks (V3)
  Global felt tiredness will be assessed using the "Fatigue Severity Scale" (FSS). The FSS is a unidimensional scale which focuses on the physical aspects of fatigue. It is a self-reported questionnaire developed to measure the impact of disabling fatigue on daily functioning. It covers several areas including physical, social, and cognitive effects. The FSS is a patient-reported outcome composed of 9-items with scores ranging from 1 = "strongly disagree" to 7 = "strongly agree".
Evaluate the feasability of measuring the impact of a personalized physical rehabilitation program at home on felt tiredness, during the program | During the two weeks of the training programm (S2 and S3)
  Tiredness felt during the training programm will be measured with the visual and analog scale for tiredness after each training session, during the two week of the program (S2 and S3).
  Score ranges from 0 to 10, 0 being "no tiredness" and 10 being "extrem tiredness"
Evaluate the feasability of measuring the impact of a personalized physical rehabilitation program at home on pain, during the program | During the two weeks of the training programm (S2 and S3)
  Pain level will be measured with the visual and analog scale for pain after each training session, during the two week of the program (S2 and S3).
  Score ranges from 0 to 10, 0 being "no pain" and 10 being "maximum thinkable pain"
Evaluate the feasability of measuring the impact of a personalized physical rehabilitation program at home on the sleep quality, in particular the duration of sleep, at S1, S2, S3 and S4 | one week before the program (S1), 2 weeks of the program (S2 and S3) and one week after the end of the program (S4)
  The duration of sleep is the total time spent spleeping. This data will be collected by the connected watch.
Evaluate the feasability of measuring the impact of a personalized physical rehabilitation program at home on the sleep quality, in particular the intensity of sleep, at S1, S2, S3 and S4 | one week before the program (S1), 2 weeks of the program (S2 and S3) and one week after the end of the program (S4)
  The intensity of sleep is the time spent in restorative phase and in slow sleep. These data will be collected by the connected watch.
Evaluate the feasability of measuring the impact of patients' satisfaction regarding the personalized physical rehabilitation program at home | 4 weeks
  Satisfaction of the patient will be assessed by a satisfaction questionnaire. Score ranges from 17 to 170, 17 being "not at all satisfied" and 170 being "totally satisfied"

CONTACTS AND LOCATIONS:
Locations (2):
- Nice CHU, Nice, Provence-Alpes-Côte d'Azur Region, France
- San Martino Hospital, Genova, Italy

IPD SHARING:
Plan to Share IPD: No